CLINICAL TRIAL: NCT03248362
Title: ELECtric Tibial Nerve Stimulation to Reduce Incontinence in Care Homes: ELECTRIC
Brief Title: ELECtric Tibial Nerve Stimulation to Reduce Incontinence in Care Homes
Acronym: ELECTRIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glasgow Caledonian University (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15/130/73
Record Dates: First submitted 2017-08-01; First posted 2017-08-14 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: A pragmatic, multicentre, placebo controlled randomised parallel group trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants & primary researchers will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPTNS Intervention (Experimental): Transcutaneous posterior tibial nerve stimulation (TPTNS) delivered in 30 minute sessions twice weekly over a 6 week period. The tibial nerve, which lies immediately posterior to the medial malleolus will be stimulated electrically using a portable TENS machine and two surface electrodes. The cathode electrode will be positioned behind the medial malleolus and the anode 10cm cephalad to it. Standardised stimulation parameters will be applied at 10 Hz frequency, 200µs-1 pulse width in continuous mode and stimulation intensity (mA-1) will be adjusted on a session-by-session basis according to individual resident comfort levels.
  Interventions: Device: Transcutaneous posterior tibial nerve stimulation
- Sham stimulation (Sham Comparator): Sham stimulation comprises low intensity, sub-clinical stimulation of the lateral sub-malleolar area, positioned specifically on the lateral aspect to avoid the tibial nerve, which runs close to the skin surface behind the medial malleolus. The stimulation parameters are identical to the TPTNS stimulation other than the intensity of the current which will be set at 4mA, rather than adjusted individually as it is in the TPTNS intervention group. The current will be initially increased until the resident reports feeling some sensation following which the current will be reduced down to 4mA. All residents will be informed that they may not feel anything with this intervention and that this is quite normal.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcutaneous posterior tibial nerve stimulation — 12 session programme (a total of 6 hours) is delivered in 30 minute sessions twice weekly over a 6 week period of tibial nerve stimulation
  Arms: TPTNS Intervention
Device: Sham stimulation — 12 session programme (a total of 6 hours) is delivered in 30 minute sessions twice weekly over a 6 week period of of the lateral sub-malleolar area
  Arms: Sham stimulation

SUMMARY:
This study aims to determine whether a programme of transcutaneous posterior tibial nerve stimulation (TPTNS) is a clinically effective treatment for urinary incontinence (UI) in care home residents and what the associated costs and consequences are.

DETAILED DESCRIPTION:
Urinary incontinence is a distressing and embarrassing condition that occurs in around 70% older people who live in nursing or residential care homes. It is common in those who have dementia as well as those with other medical conditions. Urinary incontinence has a major impact on an older person's dignity and quality of life and is linked to other health problems and relationship difficulties. It also affects a person's ability and willingness to socialise. There are not many options for treatment of urinary incontinence in older people, especially those with dementia. There are several drugs available but these can have unpleasant side-effects. Sometimes pelvic floor muscle exercises, or going to the toilet at regular intervals are tried but these can be difficult to do by those who find it hard to get around or have memory problems. They are also hard to maintain in the longer term and so older people who experience bladder leakage usually rely on the use of absorbent pads to hold the urine, rather than trying to treat the cause of the problem. Transcutaneous posterior tibial nerve stimulation (TPTNS) involves placing two sticky pads (surface electrodes) on a person's ankle and connecting these to a small, pocket sized electrical stimulator. This sends an electric pulse to the nerve near the ankle which also controls the bladder. Each treatment lasts half an hour and a total of twelve are given over a six week period. The treatment is similar to a TENS machine which is sometimes used for treating pain. It is a gentle pulsing and its strength is altered to suit the person and what is comfortable for them. TPTNS helps people with bladder leakage because it reduces the feeling of sudden urgency and the need to rush to the toilet and so gives people more warning and more time to find a toilet before they leak. TPTNS also increases the volume of urine the bladder is able to hold, so people do not need to empty their bladder as often. TPTNS has been tested in ten small studies but only one involved older people living in care homes and it only included 30 people. So far the studies have all indicated that TPTNS is safe and acceptable and that it can help bladder problems. However better quality evidence is needed that it works before it can be recommended for use in everyday treatment.

In this research the investigators will test TPTNS compared to dummy treatment in 500 people living in care homes who have urinary incontinence and who wear absorbent pads. The amount of urine they leak into participants' pads will be measured over a 24 hour period after six weeks (at the end of the TPTNS treatment programme) and after three and five months. This will tell the investigators if the treatment works and if it decreases leakage and if so, for how long. The investigators will ask the older person whether they feel their bladder leakage has changed and about any impact on their quality of life. The opinions of close family members and care home staff will be sought regarding whether they think TPTNS has had any effect on the participant. The investigators are also interested to learn about experiences of TPTNS, from residents, family and friends and all the staff involved. Costs of providing this treatment compared to the costs of providing continence care and pads will be determined and. the best ways to give TPTNS treatment in a care home, long term, will be explored with the care home staff.

ELIGIBILITY:
Inclusion Criteria:

* Care home residents:

  * with self or staff reported UI of more than once/week
  * who use the toilet or toilet aid for bladder evacuation with or without assistance
  * who wear absorbent pads to contain UI.

Exclusion Criteria:

* Care home residents:

  * with an indwelling urinary catheter
  * residents with UTI
  * residents with PVRU volume more than 300ml
  * residents with a cardiac pacemaker
  * residents with treated epilepsy
  * residents with bilateral leg ulcers
  * residents with pelvic cancer
  * residents on the palliative care register

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Volume of UI leaked | 6 weeks post randomisation.
  Volume of UI leaked over a 24 hour period

SECONDARY OUTCOMES:
Pad use | 6, 12 and 18 weeks post randomisation
  Number of pads used in 24 hours
PVRU volume | 6, 12 and 18 weeks post randomisation
  Post-void residual volume of urine scanned in bladder
PBBC | 6, 12 and 18 weeks post randomisation
  Patient Perception of Bladder Condition
FC-PBC | 6, 12 and 18 weeks post randomisation
  Family Carer Perception of Bladder Condition
S-PBC | 6, 12 and 18 weeks post randomisation
  Staff Perception of Bladder Condition
Resident DEMQOL | 6 and 18 weeks post randomisation
  Resident perception of quality of life
Staff DEMQOL | 6 and 18 weeks post randomisation
  Staff perception of quality of life
RUQ | 6 and 18 weeks post randomisation.
  Economic evaluation via a resource use questionnaire
Semi structured interviews with residents, carers and staff regarding the impact of experiences of the TPTNS intervention and any impact on quality of life | 6 and 12 weeks post randomisation
  Exploration of the experiences of the TPTNS intervention from the perspectives of residents, family carers and care home staff.
Semi-structured interviews and focus groups with care home staff and managers regarding the potential for integrating TPTNS into routine care within care homes, long-term | 6-24 weeks post randomisation
  Exploration of the factors affecting intervention implementation in the care home context and optimisation for sustainability

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Booth, Prof, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Booth J, Hagen S, McClurg D, Norton C, MacInnes C, Collins B, Donaldson C, Tolson D. A feasibility study of transcutaneous posterior tibial nerve stimulation for bladder and bowel dysfunction in elderly adults in residential care. J Am Med Dir Assoc. 2013 Apr;14(4):270-4. doi: 10.1016/j.jamda.2012.10.021. Epub 2012 Nov 30. PMID 23206722
- [Derived] Fenocchi L, Mason H, Macaulay L, O'Dolan C, Treweek S, Booth J. Cost consequence analysis of transcutaneous tibial nerve stimulation (TTNS) for urinary incontinence in care home residents alongside a randomised controlled trial. BMC Geriatr. 2023 Nov 22;23(1):766. doi: 10.1186/s12877-023-04459-z. PMID 37993786
- [Derived] Booth J, Aucott L, Cotton S, Davis B, Fenocchi L, Goodman C, Hagen S, Harari D, Lawrence M, Lowndes A, Macaulay L, MacLennan G, Mason H, McClurg D, Norrie J, Norton C, O'Dolan C, Skelton D, Surr C, Treweek S. Tibial nerve stimulation compared with sham to reduce incontinence in care home residents: ELECTRIC RCT. Health Technol Assess. 2021 Jun;25(41):1-110. doi: 10.3310/hta25410. PMID 34167637
- [Derived] Booth J, Aucott L, Cotton S, Goodman C, Hagen S, Harari D, Lawrence M, Lowndes A, Macaulay L, MacLennan G, Mason H, McClurg D, Norrie J, Norton C, O'Dolan C, Skelton DA, Surr C, Treweek S. ELECtric Tibial nerve stimulation to Reduce Incontinence in Care homes: protocol for the ELECTRIC randomised trial. Trials. 2019 Dec 16;20(1):723. doi: 10.1186/s13063-019-3723-7. PMID 31843002